CLINICAL TRIAL: NCT02912156
Title: A Randomized, Parallel, Single-Dose Study to Evaluate the Pharmacokinetics of Two Different Formulation of Voriconazole 200mg Tablets in Healthy Adult Subjects
Brief Title: Pharmacokinetics of Two Different Formulation of Voriconazole
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yung Shin Pharm. Ind. Co., Ltd. (Industry)
Collaborators: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YSP-RIH3001-01
Record Dates: First submitted 2016-09-21; First posted 2016-09-23 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Fungus Infection
Keywords: Pharmacokinetic
MeSH Terms: conditions — Mycoses | interventions — Voriconazole

ARMS (2):
- Vaway FC Tablets (Experimental): Vaway FC Tablets 200mg (Voriconazole) Dosing Regimen: Single dosing
  Interventions: Drug: Vaway FC Tablets 200mg (Voriconazole)
- VFEND FC Tablets (Active Comparator): VFEND FC Tablets 200mg (Voriconazole) Dosing Regimen: Single dosing
  Interventions: Drug: VFEND FC Tablets 200mg (Voriconazole)

INTERVENTIONS:
Drug: Vaway FC Tablets 200mg (Voriconazole)
  Arms: Vaway FC Tablets
Drug: VFEND FC Tablets 200mg (Voriconazole)
  Arms: VFEND FC Tablets

SUMMARY:
A Randomized, Parallel, Single-Dose Study to Evaluate the Pharmacokinetics of Two Different Formulation of Voriconazole 200 mg Tablets in Healthy Adult Subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult, aged between 20 to 45 years old.
2. Physically and mentally healthy subjects as confirmed by an interview, medical history review, clinical examination, laboratory tests, chest x-ray and electrocardiogram (ECG).

   * No clinically significant finding in clinical examination and laboratory tests within two months (60 days) prior to administration of study medication;
   * Normal or clinically not significant at the discretion of the investigator chest X-ray and ECG results within six months (180 days) prior to administration of study medication.
3. Body weight was above 50 kg for male and 45 kg for female.
4. The body mass index should be between 18 and 27; body mass index equals [weight (kg)]/[height (m)]2.
5. Laboratory determinations results were within normal range or considered not clinically significant by the investigator, including: Serum Glutamic Oxaloacetic Transaminase (SGOT, same as AST), Serum Glutamic Pyruvic Transaminase (SGPT, same as ALT), albumin, glucose, creatinine, uric acid, cholesterol, Triglycerides (TG), Gamma-Glutamyl-Transpeptidase (γ-GT), alkaline phosphatase, total bilirubin, Blood Urea Nitrogen(BUN),Hepatitis B surface antigen (HBsAg), Anti-Hepatitis C virus (Anti-HCV) and Anti-Human Immunodeficiency Virus (Anti-HIV) test.
6. Hematology test results were within normal range or considered not clinically significant by the investigator, including: hemoglobin, hematocrit, White Blood Cell (WBC) count, Red Blood Cell (RBC) count, platelet count and WBC count with differential.
7. Urinalysis results were within normal range or considered not clinically significant by the investigator, including: glucose, protein, RBC, WBC, epith, casts and bacteria.
8. Adequate contraceptive methods must be used during two weeks prior and two weeks after to the administration of study medication.
9. Female subject who was:

   * Using adequate contraception since last menstruation and no plan for conception during the study.
   * Non-lactating.
   * Had negative pregnancy test (urine) prior to the study.
10. Informed consent form signed.

Exclusion Criteria:

1. A history of drug or alcohol abuse within 24 weeks prior to the study.
2. History of drug allergy, allergic constitution, asthma or retinal disease.
3. Myopia worse than 6.0 diopters.
4. A clinically significant illness (such as hematological malignancy) within the past 4 weeks
5. Evidence of any clinical significant renal, cardiovascular, hepatic, hematopoietic, neurological, pulmonary or gastrointestinal disease within the past 4 weeks.
6. Planned vaccination during the study.
7. Participation of any clinical investigation during the last 60 days.
8. Regular use of any medication during the last 4 weeks.
9. Single use of any medication during the last 2 weeks.
10. Blood donation of more than 250 mL within the past 12 weeks.
11. Individuals were judged by the investigator to be undesirable as subjects.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2016-06; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration (AUC) | Plasma sample: 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 and 36 hr
Peak Drug Concentration (Cmax) | Plasma sample: 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 and 36 hr
Time to reach Cmax (Tmax) | Plasma sample: 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 and 36 hr
Elimination half-life (T1/2) | Plasma sample: 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 and 36 hr
Area under the (first) moment plasma concentration-time curve (AUMC) | Plasma sample: 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 and 36 hr

SECONDARY OUTCOMES:
Adverse events | Within 8 weeks prior to the study, subjects were screened for their eligibility.